CLINICAL TRIAL: NCT01309776
Title: Comparison of Tianeptine Versus Escitalopram for the Treatment of Depression and Cognitive Impairment in Patients With Major Depressive Disorder: A Randomized, Multicenter, Open-label Study
Brief Title: Comparison of Tianeptine Versus Escitalopram Patients Major Depressive Disorder
Acronym: CAMPION
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Bum-Hee Yu, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010-11-029
Record Dates: First submitted 2011-03-02; First posted 2011-03-07 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2013-01

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — tianeptine; Escitalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tianeptine (Experimental)
  Interventions: Drug: Tianeptine
- Escitalopram (Active Comparator)
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Tianeptine — week1 : 25mg/day q.d., week2: 37.5mg/day b.i.d. (12.5mg 1T, 12.5mg 2T
  Other Names: Stablon
  Arms: Tianeptine
Drug: Escitalopram — week1 : 5mg/day q.d., week2: 10mg/day q.d.
  Arms: Escitalopram

SUMMARY:
The primary object of this study is to confirm the superiority of tianeptine compared to escitalopram on effects that improves subjective and objective cognitive impairments in patients suffering from major depressive disorder.

DETAILED DESCRIPTION:
Along with depressive symptoms, subjective and objective cognitive impairments are frequently complained by the patients with major depressive disorder. Tianeptine acts on glutamate system and is known as a promising drug for improving cognitive impairment.

The present study aims to confirm the superiority of tianeptine compared to escitalopram on effects that improves subjective and objective cognitive impairments after a 12-week treatment in patients suffering from major depressive disorder.

ELIGIBILITY:
Inclusion Criteria:

1. Patients fulfilling DSM-IV-TR(American Psychiatric Association, 4thedition, 2000) criteria for Major Depressive Disorder diagnosis
2. The male or female patients aged more than 40 years
3. Patients able to hand in written informed consent before his/her participation in this clinical study
4. Women of childbearing potential with negative pregnancy test during screening phase and entire study period (during entire study period, able to clearly agree with effective contraception such as contraceptive pill, progesterone injection, levonorgestrel implant, estrogen ring, transdermal contraceptive agent, intra-uterine contraceptive device, sterilization operation of husband, and double contraceptive method (e.g. combination of condom, pessary, spermicide, etc. ))
5. Patients who have subjective cognitive impairment, or who have objective cognitive impairment (MMSE ≤26) without subjective cognitive impairment
6. HAM-D(17-items) total score ≥ 16

Exclusion Criteria:

1. Patients meeting more than one following patient characteristics

   1. Patients fulfilling DSM-IV-TR current or past diagnosis of any psychiatric disorders other than major depressive disorder (i.e. manic or hypomanic episode, schizophrenia, delirium, dementia, eating disorder, obsessive-compulsive disorder, panic disorder, post-traumatic stress disorder, major depressive disorder with psychotic features, mental retardation, organic brain disorder, or psychiatric disorders due to general medical condition, according to DSM-IV-TR)
   2. Patients with any substance-related disorder (excluding nicotine) within the past 12 months, as defined in DSM-IV-TR
   3. Patients with a history or presence of any neurological disorders (e.g. multiple sclerosis, seizure, etc.)
   4. Patients with any axis II disorder that prone to interfere with the evaluation of the study
2. Patients with a history or presence of any hypersensitivity to tianeptine, escitalopram or other drugs
3. Patients who receive formal psychotherapy (e.g. cognitive behavioral therapy, insight-oriented psychoanalysis, interpersonal therapy, etc.) and who have a plan for getting psychotherapy
4. Patients with any clinically significant abnormality (e.g. hepatic failure, renal failure, cardiovascular disorder, respiratory disorder, gastrointestinal disorder, endocrine disorder, neurological disorder, inflammatory disorder, neoplasm, metabolic disorder, etc.)
5. Patients who have abnormal ECG and a significant disease according to the investigator's judgment
6. Patients with any chronic liver or kidney disease
7. Patients with a family history of long QT syndrome
8. Patients previously not responders to tianeptine or escitalopram in the treatment of major depressive disorder
9. Patients who have a suicide risk according to the investigator's judgment

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2011-03; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Changes in Hamilton Rating Scale for Depression(HAM-D)score from baseline | followed up to 2,4,8,12 weeks from baseline
Changes in Korean version-California Verbal Learnign Test(K-CVLT) total score from baseline | followed up to 4,8,12 weeks from baseline
Changes in Visual Continuous Performance Test(CPT) total score from baseline | followed up to 4,8,12 weeks from baseline
Changes in Raven Progressive Matrices(RPM) total score from baseline | followed up to 4,8,12 weeks from baseline

SECONDARY OUTCOMES:
Changes in Hamilton Rating Scale for Anxiety(HAM-A) score from baseline | followed to 2,4,8,12 weeks from baseline
Changes in Clinical Clinical Global Impression- improvement(CGI-I) | followed to 2,4,8,12 weeks from baseline
Change in Response Rate from baseline | followed to 12 weeks from baseline
Change in Mini-Mental status examination(MMSE) total score from baseline | followed to 4,8,12 weeks from baseline
Change in Sexual Function Scale | followed to 2,4,8,12 weeks from baseline
Change in Clinical Global Impression- severity(CGI-S) | followed to 2,4,8,12 weeks from baseline
Change in Remission Rate from baseline | followed to 12 weeks from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Bum Hee Yu, Ph.D., Principal Investigator — Department of Pyschiatry, Sansung Medical Center
Locations (6):
- South Korea (6):
  - Inje University Paik Hospital, Goyang
  - Inje University Seoul Paik Hospital, Seoul
  - Asan Medical Center, Seoul
  - Eulji Medical College Hospital, Seoul
  - Konkuk University Medical Center, Seoul
  - Samsung Medical Center, Seoul

REFERENCES:
- [Derived] Yoo I, Woo JM, Lee SH, Fava M, Mischoulon D, Papakostas GI, Kim EJ, Chung S, Ha JH, Jeon HJ. Influence of anxiety symptoms on improvement of neurocognitive functions in patients with major depressive disorder: A 12-week, multicenter, randomized trial of tianeptine versus escitalopram, the CAMPION study. J Affect Disord. 2015 Oct 1;185:24-30. doi: 10.1016/j.jad.2015.06.038. Epub 2015 Jun 25. PMID 26142691